CLINICAL TRIAL: NCT06302907
Title: The Effect of Adding Sodium Bicarbonate 8.4% to Local Anesthesia on Pain During Upper Canine Infiltration: A Crossover Clinical Trial.
Brief Title: The Effect of Adding Sodium Bicarbonate 8.4% to Local Anesthesia on Pain During Upper Canine Infiltration
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Wataniya University (Other)
Responsible Party: Principal Investigator, Tarek Khaled Abou Agwa, Senior lecturer, Al-Wataniya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M/45- 14.1.2023
Record Dates: First submitted 2024-03-01; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Local Anesthetic Complication
Keywords: Upper canine infiltration; Lidocaine; Sodium bicarbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buffered LA (Active Comparator): AA buffered 2% lidocaine with 1:80000 epinephrine and sodium bicarbonate 8.4% was used for one site
  Interventions: Procedure: Buffered Local anaesthesia; Procedure: Unbuffered Local anaesthesia
- Unbuffered LA (Active Comparator): an unbuffered 2% lidocaine with 1: 80000 epinephrine for the other site at the same appointment.
  Interventions: Procedure: Buffered Local anaesthesia; Procedure: Unbuffered Local anaesthesia

INTERVENTIONS:
Procedure: Buffered Local anaesthesia — A buffered 2% lidocaine with 1:80000 epinephrine and sodium bicarbonate 8.4% was used for one site
Procedure: Unbuffered Local anaesthesia — an unbuffered 2% lidocaine with 1: 80000 epinephrine for the other site at the same appointment.

SUMMARY:
The aim of the present study was to evaluate the pain during local anesthetic buccal infiltration for the maxillary canines after adding Sodium Bicarbonate 8.4% during local anesthesia.

DETAILED DESCRIPTION:
Materials and Methods The present research was approved by the Institutional Review Board of the College of Dentistry at Al Wataniya Private University (M/45- 14.1.2023).

30 healthy patients were recruited, aged between 15-50 years, and divided into two groups (15 males and 15 females). Every patient had to meet the following conditions:

* Caries free with no restorations, periapical lesions, or history of trauma at the site of injection.
* Willingness to participate in the study and ability to describe and evaluate their pain.
* No painkillers, or sedatives taken for at least 24 hours so that pain assessment isn't affected.
* No allergy to local anesthetics.
* No pregnancy. Each patient received buccal infiltration with the anesthetic solution alone at one upper canine site and local anesthetic with added sodium bicarbonate at the other site. The local anesthetic used was 2% Lidocaine with 1:80.000 Epinephrine produced by New-Stetic S.A.- Colombia. Whereas 8.4% Bicarbonate Sodium was produced by TCE - UK. Injections were performed using 25 mm short needles (Gauge 27) manufactured by C-K Dental - South Korea.

Consent for each patient was obtained before the clinical session. Local infiltration was performed using a one-third cartridge (0.6 mL) of the local anesthetic on one side and local anesthetic with added Sodium Bicarbonate on the counterpart side leaving 5 minutes between the injections.

Alkalinization of the local anesthetic was performed using the technique described by Saatchi et al13. 0.2 mL of the anesthetic solution was extracted using a tuberculin syringe and then discarded. 0.2 mL sodium bicarbonate was then loaded and added to the cartridge. Afterward, the solution was slowly shaken 20 times and ready to be administered with a cartridge syringe.

The 100 mm Visual Analog Scale VAS was utilized as the most commonly used assessment tool to determine the severity of the pain14 where 0 indicates that the patient does not feel pain, while 10 points to unbearable severe pain. The patients must rely on their own experience to confirm the pain's severity.

ELIGIBILITY:
Inclusion Criteria:

* Caries free with no restorations, periapical lesions, or history of trauma at the site of injection.
* Willingness to participate in the study and ability to describe and evaluate their pain.
* No painkillers, or sedatives taken for at least 24 hours so that pain assessment isn't affected.

Exclusion Criteria:

* allergy to local anesthetics.
* pregnancy

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain on injection | one week
  - Pain was measured on a visual analogue scale (VAS) starting from 0 which represents (no pain at all) and ending with 10 which represents (the most severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Tarek A Agwa, Senior Lect, Principal Investigator — Al Wataniya Private University
Locations (1):
- Al Wataniya Private University, Hama, Hama Government, Syria

IPD SHARING:
Plan to Share IPD: No